CLINICAL TRIAL: NCT02206607
Title: A Phase 1, Randomized, Open-label, Cross-over, Single-day Study Of Pf-04937319 To Characterize Relative Bioavailability, Tolerability, And Pharmacodynamics Of Four Oral Formulations In Adults With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: Study To Compare Single Dose Of Three Modified Release Formulations Of PF-04937319 With Immediate Release Material-Sparing-Tablet (IR MST) Formulation Previously Studied In Adults With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1621015
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Phase 1; bioavailability; type 2 diabetes mellitus; PF-04937319
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04937319 IR MST (Experimental): Reference formulation
  Interventions: Drug: PF-04937319 IR MST
- PF-04937319 MR 1 (Experimental): Test MR #1
  Interventions: Drug: PF-04937319 MR 1
- PF-04937319 MR 2 (Experimental): Test MR #2
  Interventions: Drug: PF-04937319 MR 2
- PF-04937319 MR 3 (Experimental): Test MR #3
  Interventions: Drug: PF-04937319 MR 3

INTERVENTIONS:
Drug: PF-04937319 IR MST — Immediate release material sparing tablet (IR MST) administered as 150 mg with morning meal and 100 mg with lunch
  Arms: PF-04937319 IR MST
Drug: PF-04937319 MR 1 — Modified release formulation #1 administered with the morning meal at a dose predicted to yield exposure (AUC24) equivalent to 300 mg IR MST
  Arms: PF-04937319 MR 1
Drug: PF-04937319 MR 2 — Modified release formulation #2 administered with the morning meal at a dose predicted to yield exposure (AUC24) equivalent to 300 mg IR MST
  Arms: PF-04937319 MR 2
Drug: PF-04937319 MR 3 — Modified release formulation #3 administered with the morning meal at a dose predicted to yield exposure (AUC24) equivalent to 300 mg IR MST
  Arms: PF-04937319 MR 3

SUMMARY:
Study B1621015 will characterize bioavailability, tolerability and pharmacodynamics of three modified release formulations of PF-04937319 compared with the immediate release material-sparing-tablet (IR MST) formulation in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 2 diabetes, on stable background metformin therapy either alone or in combination with another oral anti-diabetic agent (OAD) excluding thiazolidinediones (TZDs)

Exclusion Criteria:

* Patients with cardiovascular event within 6 months of screening
* Patients with diabetic complications
* Female subjects who are pregnant or planning to become pregnant
* Subjects with unstable medical conditions (eg, hypertension)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - High Point Clinical Trials Center, High Point, North Carolina
  - Clinical Trials of Texas, Inc., San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to being enrolled in the 4 period crossover, participants were required to complete an open-label, sponsor-provided metformin period. 42 participants started the metformin period and of those 42 participants, 39 were enrolled in the 4 period crossover and received at least 1 dose PF-04937319.
Groups:
- Metformin Run-In: Participants received open-label, sponsor-provided metformin tablet(s) orally at a dose in multiples of 500 mg (minimum dose 500 mg, maximum dose 2500 mg). Participants who met eligibility criteria on metformin were then randomized to 1 of 4 treatment sequences.
- Sequence ADBC: PF-04937319 150+100 mg IR First: Participants received immediate-release material sparing tablet (IR MST) administered orally at 150 mg with morning meal and 100 mg with lunch, followed by PF-04937319 modified-release formulation #3 (MR3) 330 mg, followed by PF-04937319 modified-release formulation #1 (MR1) 250 mg, followed by PF-04937319 modified-release formulation #2 (MR2) 300 mg. There was a 5 to 10-day washout between dosing across the 4 regimens.
- Sequence BACD: PF-04937319 250 mg MR1 First: Participants received PF-04937319 MR1 250 mg, followed by PF-04937319 150+100 mg IR, followed by PF-04937319 300 mg MR2, followed by PF-04937319 330 mg MR3. There was a 5 to 10-day washout between dosing across the 4 regimens.
- Sequence CBDA: PF-04937319 300 mg MR2 First: Participants received PF-04937319 300 mg MR2, followed by PF-04937319 250 mg MR1, followed by PF-04937319 330 mg MR3, followed by PF-04937319 150+100 mg IR. There was a 5 to 10-day washout between dosing across the 4 regimens.
- Sequence DCAB: PF-04937319 330 mg MR3 First: Participants received PF-04937319 330 mg MR3, followed by PF-04937319 300 mg MR2, followed by PF-04937319 150+100 mg IR, followed by PF-04937319 250 mg MR1. There was a 5 to 10-day washout between dosing across the 4 regimens.
Period: Open-Label Run-In
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 42 | 0 | 0 | 0 | 0
Completed | 39 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0
Period: First Intervention Period
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 11 | 10
Completed | 0 | 9 | 9 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: First Washout Period 5 to 10 Days
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 11 | 10
Completed | 0 | 9 | 9 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 11 | 10
Completed | 0 | 9 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Insufficient Clinical Response | 0 | 0 | 0 | 1 | 0
Period: Second Washout Period 5 to 10 Days
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 10 | 10
Completed | 0 | 9 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 10 | 10
Completed | 0 | 9 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Third Washout Period 5 to 10 Days
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 10 | 10
Completed | 0 | 9 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Metformin Run-In | Sequence ADBC: PF-04937319 150+100 mg IR First | Sequence BACD: PF-04937319 250 mg MR1 First | Sequence CBDA: PF-04937319 300 mg MR2 First | Sequence DCAB: PF-04937319 330 mg MR3 First
Started | 0 | 9 | 9 | 10 | 10
Completed | 0 | 9 | 9 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who received at least 1 dose of study treatment (PF-04937319).
Groups:
- All Participants: Participants received at least 1 dose of PF-04937319.
Arm/Group | All Participants
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf]
Description: AUCinf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time.
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: The pharmacokinetic (PK) parameter analysis population included all randomized participants who received at least 1 dose of PF-04937319 and who had at least 1 of the PK parameters of interest measured and available in at least 1 period; number of participants analyzed (N) is number of evaluable participants for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- PF-04937319 150+100 mg IR: Participants received immediate-release material sparing tablet (IR MST) administered orally at 150 mg with morning meal and 100 mg with lunch. There was a 5 to 10-day washout between dosing across the 4 regimens.
- PF-04937319 250 mg MR1: Participants received modified-release formulation #1 administered orally at 250 mg tablet with morning meal. There was a 5 to 10-day washout between dosing across the 4 regimens.
- PF-04937319 300 mg MR2: Participants received modified-release formulation#2 administered orally at 300 mg with morning meal. There was a 5 to 10-day washout between dosing across the 4 regimens.
- PF-04937319 330 mg MR3: Participants received modified-release formulation#3 administered orally at 330 mg with morning meal. There was a 5 to 10-day washout between dosing across the 4 regimens.
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 31 | 37 | 36
nanogram*hour/milliliter (ng*hr/mL) | 10690 (26) | 3187 (59) | 2725 (35) | 3430 (37)
Statistical Analysis 1: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 250 mg MR1; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR1/IR = 31.27, 90% CI 2-sided [28.09 to 34.80]
Statistical Analysis 2: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 300 mg MR2; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR2/IR = 25.56, 90% CI 2-sided [23.11 to 28.27]
Statistical Analysis 3: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 330 mg MR3; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR3/IR = 32.04, 90% CI 2-sided [28.93 to 35.49]

2. Primary Outcome: Change From Reference in Weighted-Mean-Daily-Glucose (WMDG) on Day 1
Description: MWG was calculated as the area under the curve (AUC) for the full 24 hours expressed.
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, and 24 hours post-dose
Population: The pharmacodynamic analysis included participants who had taken at least 1 dose of PF-04937319 and who had WMDG assessment for at least 1 modified-release formulation and the Reference (IR MST) formulation; n=number of participants evaluated in respective arms for category.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 36 | 36 | 36 | 36
milligrams per deciliter (mg/dL)
  Observed (n=36,33,32,35) | 159.47 (42.949) | 176.24 (42.648) | 170.85 (38.928) | 180.47 (50.099)
  Change From Reference (36,33,32,35) | NA (NA) — No measure type or method of dispersion was calculated, as the 'PF-04937319 150+100 mg IR' arm is the Reference. | 15.55 (19.358) | 15.96 (17.122) | 20.15 (20.005)
Statistical Analysis 1: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 250 mg MR1; Test type: Superiority or Other; p = 1.0000, Mixed Models Analysis — 1-sided p-value; Treatment, period, sequence as fixed effects and subjects-within-sequence as random effects; Least Square Mean = 15.72, 80% CI 2-sided [11.39 to 20.06], Standard Error of Mean 3.357
Statistical Analysis 2: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 300 mg MR2; Test type: Superiority or Other; p = 1.000, Mixed Models Analysis — 1-sided p-value; Treatment, period, sequence as fixed effects and subjects-within-sequence as random effects; Least Square Mean = 16.31, 80% CI 2-sided [11.93 to 20.70], Standard Error of Mean 3.399
Statistical Analysis 3: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 330 mg MR3; Test type: Superiority or Other; p = 1.0000, Mixed Models Analysis — 1-sided p-value; Least Square Mean = 20.38, 80% CI 2-sided [16.13 to 24.62], Standard Error of Mean 3.291

3. Secondary Outcome: Maximum Observed PF-04937319 Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: The PK parameter analysis population included all randomized participants who received at least 1 dose of PF-04937319 and who had at least 1 of the PK parameters of interest measured and available in at least 1 period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
ng/mL | 641.2 (22) | 161.8 (37) | 171.3 (24) | 236.2 (24)
Statistical Analysis 1: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 250 mg MR1; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR1/IR = 25.21, 90% CI 2-sided [23.28 to 27.31]
Statistical Analysis 2: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 300 mg MR2; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR2/IR = 26.38, 90% CI 2-sided [24.36 to 28.57]
Statistical Analysis 3: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 330 mg MR3; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR3/IR = 36.94, 90% CI 2-sided [34.09 to 40.02]

4. Secondary Outcome: PF-04937319 Plasma Concentration at 5 Hours After Morning Dose (C5)
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
ng/mL | 413.2 (26) | 124.3 (43) | 154.3 (29) | 202.1 (30)

5. Secondary Outcome: PF-04937319 Plasma Concentration at 16 Hours After Morning Dose (C16)
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
ng/mL | 324.7 (34) | 74.49 (57) | 58.88 (37) | 77.92 (37)

6. Secondary Outcome: PF-04937319 Plasma Concentration at 24 Hours After Morning Dose (C24)
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
ng/dL | 171.1 (37) | 56.04 (64) | 39.38 (52) | 48.17 (47)

7. Secondary Outcome: Ratio of Maximum to Approximate Trough PF-04937319 Concentration (Cmax/C24)
Description: Cmax/C24 is the ratio of maximum to approximate trough concentration, where Cmax is the overall maximum observed plasma concentration and C24 is the plasma concentration at 24 hours after the morning dose.
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
ratio | 3.748 (33) | 2.887 (49) | 4.350 (48) | 4.903 (43)

8. Secondary Outcome: Time to Reach Maximum Observed PF-04937319 Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
hours | 8.00 [3.00 to 15.2] | 6.00 [4.00 to 48.0] | 5.00 [1.00 to 7.07] | 5.00 [3.00 to 7.00]

9. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable PF-04937319 Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 39 | 39 | 38
ng*hr/mL | 10560 (26) | 3287 (55) | 2644 (34) | 3369 (34)
Statistical Analysis 1: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 250 mg MR1; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR1/IR = 31.06, 90% CI 2-sided [28.28 to 34.10]
Statistical Analysis 2: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 300 mg MR2; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR2/IR = 24.96, 90% CI 2-sided [22.73 to 27.40]
Statistical Analysis 3: Comparison: PF-04937319 150+100 mg IR vs PF-04937319 330 mg MR3; Test type: Superiority or Other; Adjusted Geometric Mean Ratio MR3/IR = 31.69, 90% CI 2-sided [28.86 to 34.81]

10. Secondary Outcome: Terminal Elimination Half-Life (t1/2)
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 11, 12.5, 14, 16, 20, 24, 36, 48, and 72 hours post-dose
Population: The PK parameter analysis population included all randomized participants who received at least 1 dose of PF-04937319 and who had at least 1 of the PK parameters of interest measured and available in at least 1 period; number of participants analyzed (N) is number of evaluable participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 38 | 31 | 37 | 36
hour | 8.648 (2.7801) | 12.10 (5.5922) | 13.52 (6.9657) | 12.62 (6.1783)

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last study drug administration in Period 4
Population: The safety analysis population included all participants who received at least 1 dose of open-label, sponsor-provided metformin.
Measure: Number; unit: participants
Groups:
- Metformin Run-In: Participants received open-label, sponsor-provided metformin tablet(s) orally at a dose in multiples of 500 mg (minimum dose 500 mg, maximum dose 2500 mg). Participants who met eligibility criteria on metformin were then randomized to 1 of 4 treatment regimens.
Arm/Group | Metformin Run-In | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Number analyzed (Participants) | 42 | 38 | 39 | 39 | 38
participants
  AEs | 2 | 16 | 11 | 16 | 10
  SAEs | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration in Period 4
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Metformin Run-In | PF-04937319 150+100 mg IR | PF-04937319 250 mg MR1 | PF-04937319 300 mg MR2 | PF-04937319 330 mg MR3
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38 | 0/39 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 1/42 | 11/38 | 6/39 | 10/39 | 5/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin Run-In (N=42) | PF-04937319 150+100 mg IR (N=38) | PF-04937319 250 mg MR1 (N=39) | PF-04937319 300 mg MR2 (N=39) | PF-04937319 330 mg MR3 (N=38)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Toothache (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 7 | 2 | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.